CLINICAL TRIAL: NCT04573127
Title: Epidemiological Characteristics of the Population of Persons With Gender Dysphoria : Data From the Cohort Follow-up in CHRU de Nancy
Brief Title: Gender Dysphoria: Epidemiological Data
Acronym: DyGenEpi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI159
Record Dates: First submitted 2020-08-07; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive study — Retrospective analysis of existing data collected as a part of the regular follow-up
  Other Names: Retrospective analysis of existing data collected as a part of the regular follow-up

SUMMARY:
Retrospective study in a single academic regional transgender referral center. data from the cohort follow-up in CHRU de Nancy

ELIGIBILITY:
Retrospective analysis of available data as a part of the regular care of subjects with gender dysphoria. All measurements were made at the time of the routine follow-up visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the outpatient clinic at our department of endocrinology
Study Population: Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the outpatient clinic at our department of endocrinology
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Incdience rate of cardiovascular diseases | 2004-2020
  Number of new cases of arterial hypertension, stroke, myocardial infarction during the specified period (2004-2020) /Time each person was observed, totaled for all persons
Incidence rate of dyslipidemia | 2004-2020
  Number of new cases of dyslipidemia during the specified period (2004-2020) /Time each person was observed, totaled for all persons

SECONDARY OUTCOMES:
Incidence rate of oncological diseases | 2004-2020
  Number of new cases of malignancies during the specified period (2004-2020) /Time each person was observed, totaled for all persons
Incidence rate of psychiatric diseases | 2004-2020
  Number of new cases of psychiatric diseases malignancies during the specified period (2004-2020) /Time each person was observed, totaled for all persons
Overall mortality rate | 2004-2020
  Mortality during the specified period (2004-2020) /Time each person was observed, totaled for all persons

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided